CLINICAL TRIAL: NCT03174548
Title: A Phase 1, Randomized, Single-center, Open-label, Three-sequence, Three-period, Three-treatment Crossover Study to Evaluate the Effect of Food on the Single-dose Pharmacokinetics of Sotagliflozin and to Explore the Relative Bioavailability of Sotagliflozin Oral Tablet to Oral Solution in Healthy Male and Female Subjects
Brief Title: A Study to Evaluate the Effect of Food on the Pharmacokinetics of Sotagliflozin and to Explore the Relative Bioavailability in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PKM15047; 2016-004650-15 (EudraCT Number); U1111-1189-5094 (Other: UTN)
Record Dates: First submitted 2017-05-31; First posted 2017-06-02 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Fed Tablet period (Test, T) (Experimental): Sotagliflozin oral in fed conditions
  Interventions: Drug: Sotagliflozin (SAR439954)
- Fasted Tablet period (Reference, R) (Experimental): Sotagliflozin oral in fasting conditions
  Interventions: Drug: Sotagliflozin (SAR439954)
- Oral Solution period (S) (Experimental): Sotagliflozin oral solution in fasting conditions
  Interventions: Drug: Sotagliflozin (SAR439954)

INTERVENTIONS:
Drug: Sotagliflozin (SAR439954) — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: Fasted Tablet period (Reference, R); Fed Tablet period (Test, T)
Drug: Sotagliflozin (SAR439954) — Pharmaceutical form: solution
  Route of administration: oral
  Arms: Oral Solution period (S)

SUMMARY:
Primary Objective:

To evaluate the effect of food on the single-dose pharmacokinetics of sotagliflozin relative to a fasted state in healthy adult male and female subjects.

Secondary Objectives:

* To evaluate the effect of food on the single-dose pharmacokinetics of the main metabolite (sotagliflozin 3-O-glucuronide) relative to a fasted state in healthy adult male and female subjects.
* To investigate the relative bioavailability of sotagliflozin tablet to oral solution under fasting conditions
* To evaluate safety and tolerability of single-dose sotagliflozin under fed and fasted conditions in healthy adult male and female subjects.

DETAILED DESCRIPTION:
The study duration per subject will be 26 to 83 days and will consist of a screening period of 2-28 days, a treatment period of 6 days each for Periods 1, 2 and 3, a washout between treatment periods of 1-14 days, and follow up visit 10-15 days after the last Investigational Medicinal Product administration in period 3.

ELIGIBILITY:
Inclusion criteria :

* Healthy male and female subjects, between 18 and 55 years of age, inclusive, at the time of screening.
* Body weight between 50.0 and 100.0 kg, inclusive, if male, and between 40.0 and 90.0 kg, inclusive, if female; body mass index between 18.0 and 30.0 kg/m2, inclusive.
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination), vital signs, ECG, and clinical laboratory parameters.

Exclusion criteria:

* Any history or presence of clinically relevant illness at screening, which could interfere with the objectives of the study or the safety of the subject's participation.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month).
* Blood donation any volume, within 2 months before inclusion.
* Symptomatic postural hypotension.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
* History or presence of drug or alcohol abuse.
* Smoking more than 5 cigarettes or equivalent per day, unable to stop smoking during the study.
* If female, pregnancy, breast-feeding.
* Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication; any vaccination within the last 28 days and any biologics (antibody or its derivatives) given within 4 months before inclusion.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Maximum plasma drug concentration (Cmax) of sotagliflozin | From 0 to 120 hours after sotagliflozin intake
Area under curve (AUC) of sotagliflozin | From 0 to 120 hours after sotagliflozin intake

SECONDARY OUTCOMES:
Sotagliflozin (tablet and oral solution):Apparent volume of distribution during terminal phase after non-intravenous administration (Vz/F) | From 0 to 120 hours after sotagliflozin intake
Sotagliflozin (tablet and oral solution): Time to reach maximum plasma concentration (tmax) | From 0 to 120 hours after sotagliflozin intake
Sotagliflozin (tablet and oral solution): Elimination half-life (t1/2z) | From 0 to 120 hours after sotagliflozin intake
Sotagliflozin-O-glucuronide (tablet and oral solution): Cmax | From 0 to 120 hours after sotagliflozin intake
Sotagliflozin-O-glucuronide (tablet and oral solution): tmax | From 0 to 120 hours after sotagliflozin intake
Sotagliflozin-O-glucuronide (tablet and oral solution): t1/2z | From 0 to 120 hours after sotagliflozin intake
Sotagliflozin-O-glucuronide (tablet and oral solution): Area under the plasma concentration-time curve from time zero to time of last measurable concentration (AUClast) | From 0 to 120 hours after sotagliflozin intake
Sotagliflozin-O-glucuronide (tablet and oral solution): AUC | From 0 to 120 hours after sotagliflozin intake
Relative bioavailability (Frel) | From 0 to 120 hours after sotagliflozin intake
Number (%) of subjects with treatment emergent adverse events | Over 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 826001, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org